CLINICAL TRIAL: NCT06743607
Title: Spinal Stimulation to Improve Upper Extremity Recovery in the Home (SSTIM UE Recover [SURe])
Brief Title: Spinal Stimulation for Upper Extremity Recovery in the Home
Acronym: SURe
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Hospital (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Candace Tefertiller, Executive Director of Research and Evaluation, Craig Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2274573-1
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-12

CONDITIONS: Cervical Spinal Cord Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Active Comparator): For the immediate intervention group, each participant will complete the following:
  * Initial baseline evaluation
  * 24 training sessions (3x/week for eight weeks) of UE Functional Task Practice (FTP)+TSS (two training sessions/week will be completed in the home with caregiver/companion support; the third weekly session will be conducted via videoconference with a research therapist)
  * Post-treatment evaluation (after eight weeks of training) and follow-up evaluation (four weeks after post-treatment evaluation).
  * Post-treatment and follow-up assessments will be conducted over two days: assessments completed without TSS on day one and with TSS on day two.
  Interventions: Behavioral: Immediate Intervention
- Waitlist Control (Active Comparator): The waitlist control group will participate in a protocol similar to the immediate intervention group, except:
  * 12-week waiting period before starting the active intervention.
  * Assessments will be completed at 0, 8, and 12 weeks before starting the active intervention to control for spontaneous recovery.
  * Post-treatment evaluation (after eight weeks of training)
  * Follow-up assessment (four weeks after the post-treatment evaluation).
  Interventions: Behavioral: Waitlist control

INTERVENTIONS:
Behavioral: Immediate Intervention — Participants will engage in a home exercise therapy program in combination with transcutaneous spinal stimulation intended to focus on the upper extremities that commences immediately after enrollment.
  Arms: Immediate Intervention
Behavioral: Waitlist control — Participants will engage in a home exercise therapy program in combination with transcutaneous spinal stimulation intended to focus on the upper extremities that commences 12 weeks after enrollment.
  Arms: Waitlist Control

SUMMARY:
The purpose of this research is to evaluate the safety, feasibility, and tolerability of non-invasive spinal stimulation used in the home and/or community in combination with a functional home exercise program for the upper extremities (arm/hand function) as well as their combined impacts on changes in upper extremity function. The expected duration of participation in this study is about 31-33 hours over a 13-25-week period. Enrollees in this study will be randomly assigned to one of two groups: 1) upper extremity functional task-specific training combined with non-invasive transcutaneous spinal stimulation, or 2) waitlist control, which involves the same intervention, but with a 12-week delayed start. Participants complete initial testing (one time if in group one and three times [at weeks 0, 8, and 12] if in group two), 24 1-hour training sessions (2x/week in home with caregiver/companion support and 1x/week with research team in person or via video conference for 8 weeks), a post-treatment evaluation, and a final evaluation (4 weeks after post-treatment).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* History of traumatic SCI
* Less than 12 months post SCI
* SCI injury level C1-C8
* SCI categorized as AIS B-D
* Have passive range of motion (ROM) within functional limits at wrists, shoulders, and elbows
* Have caregiver support to attend three in-person sessions and ongoing training at home
* Have a caregiver who, in the judgment of the research team, is qualified to assist the participant in the safe use of TSS
* Able to complete in-person training sessions and return to Craig Hospital for assessments
* Experience no complicating physical or cognitive conditions as determined by their physician that would preclude the safe use of electrical stimulation
* If using prescribed anti-spasticity medications, must be at a stable dose for at least four weeks prior to starting study procedures
* Agrees to comply with investigational devices instructions for use, protocol visits, and return of the device
* Able to provide informed consent

Exclusion Criteria:

* Experience unstable chronic cardiac or respiratory complaints
* Have a recent history of fracture, contractures, or skin pressure injuries that might interfere with the intervention
* Received Botox injections to the UEs, neck, or hands within the last three months
* Pregnant, planning to become pregnant, or currently breastfeeding
* Have breakdown in skin area that will come into contact with electrodes
* Prior nerve or tendon transfer procedure for the UEs
* Concurrently are participating in another drug or device trial that may interfere with this study
* Have an implanted pacemaker, spinal cord stimulator, ventriculoperitoneal shunt, deep brain stimulator, or intrathecal pump
* In the opinion of the investigators, the study is not safe or appropriate for the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Capabilities of Upper Extremity Questionnaire (CUE-Q) | Weeks 0, 8, 12, 21, and 25
  The CUE-Q version 2.1 measures functional limitation and perceived difficulty of performing actions with upper extremities in individuals with tetraplegia. The CUE-Q has 32 items; each scored on a 1-to-7-point scale representing self-perceived difficulty with total scores ranging from 32 to 224 (higher scores demonstrating greater UE function) and right and left scores assessed separately

SECONDARY OUTCOMES:
Graded Refined Assessment of Strength, Sensibility, and Prehension (GRASSP) | Weeks 0, 8, 12, 21, and 25
  This multimodal test measures sensorimotor and prehension function in three domains important in describing arm and hand function
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) | Weeks 0, 8, 12, 21, and 25
  The ISNCSCI is a universal classification tool for SCI based on a standardized sensory and motor exam. The ISNCSCI involves a detailed examination to determine the sensory and motor levels for both the right and left sides, the overall neurological level of the injury, and the completeness of the injury as designated by the American Spinal Cord Injury Association (ASIA) Impairment Scale (AIS). The motor exam also results in a total Upper Extremity Motor Score (UEMS) ranging from 0 to 50, with higher scores indicative of greater UE strength.
Pinch and Grasp Force | Weeks 0, 8, 12, 21, and 25
  Pinch and grasp force will be measured by the Commander Echo Console with the JTech Pinch and Hand Dynamometer to quantify finger and grasp strength.
Global Rating of Change (GRC) | Weeks 8, 12, 21, and 25
  The GRC assesses perceived change from an intervention. The scale is designed to quantify an individual's perceived improvement or deterioration over time. The magnitude of the change is then scored on a visual analog scale. GRC scales have been recommended for use as a core outcome measure in rehabilitation studies to improve the applicability of information from clinical trials to clinical practice.
Satisfaction with Treatment Scale | Weeks 8, 12, 21, and 25
  The Satisfaction with Treatment Scale is a 6-point scale (0=strongly disagree; 5= strongly agree) used to rate satisfaction with treatment in previous intervention studies conducted in the home environment85 and will be modified specifically to address the transcutaneous spinal stimulation (TSS) intervention.
Qualitative Questions | Weeks 8 and 21
  Participants and caregivers will be asked questions regarding their experience during the intervention, such as their likes and dislikes, notable changes or observations, and overall satisfaction with using TSS in their homes
Canadian Occupational Performance Measure (COPM) | Weeks 0, 8, 12, 21, and 25
  The COPM is an individualized, client-centered instrument designed to measure an individual's self-perception of physical functioning and satisfaction in the activities identified as important by the client. The COPM will directly assess the true importance of functional improvements with regard to the subject's ability to perform activities of daily living and/or to function occupationally.
International Spinal Cord Injury Quality of Life Basic Data Set (QoL-BDS) Version 2.0 | Weeks 0, 8, 12, 21, and 25
  This instrument measures self-reported quality of life across four domains: overall well-being, physical health, psychological health, and social life. For each domain, respondents are asked to rate their satisfaction on a 0-10 scale (0=completely dissatisfied; 10=completely satisfied).
International Spinal Cord Injury Pain Basic Data Set (ISCIPBDS) Version 3.0 | Weeks 0, 8, 12, 21, and 25
  This instrument identifies pain region, pain type (e.g., nociceptive, neuropathic), and treatments used to reduce pain in addition to pain intensity on a 0-10 scale (0=no pain; 10=pain as bad as you can imagine) and interference with various aspects of the respondent's life on a 0-10 scale (0=no interference; 10=extreme interference).

OTHER OUTCOMES:
Demographic Information | Week 0
  Demographic information will include: age, sex, race/ethnic background, pre-injury education, employment status, marital status, and living situation.
Injury Characteristics | Week 0
  Injury information will include: date of injury, cause of injury, baseline AIS classification, and injury level.

CONTACTS AND LOCATIONS:
Locations (1):
- Craig Hospital, Englewood, Colorado, United States